CLINICAL TRIAL: NCT06604299
Title: Digital Mindfulness Meditation-enhanced Cognitive Behavioral Therapy (CBT-MM) for Binge Eating Disorder User-Testing
Brief Title: Digital Mindfulness Meditation-enhanced Cognitive Behavioral Therapy (CBT-MM) for Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeshiva University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 127265; K23AT012126 (NIH)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Binge Eating Disorder
Keywords: binge eating; eating disorders; obesity
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital CBT-MM (Experimental): Digital CBT-MM is a digital intervention including mindfulness and cognitive behavioral elements for individuals with binge eating disorder. Mindful Courage will consist of 18-weeks of self-guided modules. Elements included in the intervention include psychoeducation, self-monitoring, regular eating, goal-setting, weekly weighing, eating a sufficient amount of food at each meal, eating a range of foods (including foods that patients may fear), reduction of overvaluation of weight and shape, addressing shape/body checking or avoidance, behavior chain analysis, problem solving, awareness and acceptance of binge eating urges, thoughts and emotions, values awareness, values clarification, values-based decision making, self-compassion, exploring needs underlying binge eating urges, mindful eating, hunger and fullness awareness, self-compassion, and self-care. Weekly mindfulness practice (at least 3x per week) is heavily emphasized.
  Interventions: Behavioral: Meditation-enhanced Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Meditation-enhanced Cognitive Behavioral Therapy — Self-guided online intervention

SUMMARY:
The investigators will evaluate the acceptability and feasibility of a 18-week long digital mindfulness-based and cognitive behavioral therapy intervention for binge eating disorder.

This study is a prospective single-arm trial during the intervention development phase. Following this phase, after the intervention has been further developed, a subsequent study (with a different clinicaltrials.gov identification #) will utilize a randomized control trial design.

DETAILED DESCRIPTION:
Procedures include completing: (1) pre-intervention screening assessment; (2) an initial baseline visit; (3) 18-week web-based intervention; and (4) a post-intervention assessment (18-weeks after baseline).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Meeting DSM-5 criteria for Binge Eating Disorder (BED)
* English-speaking

Exclusion Criteria:

* BMI < 18.5
* Requiring immediate treatment for medical complications
* Current anorexia or bulimia nervosa or purging behaviors within the past year
* Already receiving treatment for an ED or participating in a weight loss program or psychotherapy focused on weight (psychotherapy for other conditions was allowed)
* Currently pregnant or breast-feeding
* Experiencing other severe psychopathology or medical illness that would limit the participants' ability to comply with the demands of the current study (e.g. active psychotic disorder, cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Acceptability | 18-week treatment period
  Single-items measuring dimensions of acceptability, including overall satisfaction, engagement, visual appeal of content, understandability of program material, desire to continue the program, and overall helpfulness. Scores for each item range from 1 to 5, , with higher scores indicating better acceptability.
Feasibility/Completion | 18-week treatment period
  Module completion, ranging from 0 to 100%

SECONDARY OUTCOMES:
Changes in Emotion Dysregulation | Baseline to post-treatment (18-weeks)
  Difficulties in Emotion Regulation Short Form (DERS-SF). Total scores are the average of each of the subscales, and range from 1 to 5. Higher scores indicate more emotion dysregulation
Changes in Mindfulness | Baseline to post-treatment (18-weeks)
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Total scores range from 0 to 40, with higher scores indicating greater mindfulness.
Changes in Objective Binge Eating Episodes | Baseline to post-treatment (18-weeks)
  Eating Disorder Examination-Questionnaire (EDE-Q). The EDE-Q asks participants to report on the number of episodes in the last 28 days in which they ate a large amount of food with a sense of loss of control.
Change in Body Mass Index (BMI) | Baseline to post-treatment (18-weeks)
  Computed using self-reported height and body weight
Changes in Dietary Restraint | Baseline to post-treatment (18-weeks)
  Dietary restraint subscale of the EDE-Q (EDE-Q; Fairburn & Beglin, 1994). Scores range from 0 to 6, and higher scores indicate higher restraint.
Changes in Quality of Life | Baseline to post-treatment (18-weeks)
  Eating Disorder Quality of Life scale (EDQOL; Engel et al., 1996). Scores on each item range from 1 to 4, with higher scores indicating better quality of life.
Changes in Depression Symptoms | Baseline to post-treatment (18-weeks)
  Beck Depression Inventory-II (BDI-II; Beck et al., 1996). Scores range from 0 to 63, with higher scores indicating higher depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeshiva University, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No